CLINICAL TRIAL: NCT06531356
Title: Efficiency of Autologous Amniotic Fluid Injection in the Healing of Cesarean Section Scar in High-Risk Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Hend Mahmoud Abdelghany, Lecturer of Obstetrics and Gynecology, Cairo University, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS-141-2023
Record Dates: First submitted 2024-02-13; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: High Risk Pregnancy; Healing Surgical Wounds
Keywords: amniotic fluid; cesarean section scar (healing)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases (Experimental)
  Interventions: Biological: autologous amniotic fluid
- control (Active Comparator)
  Interventions: Other: No amniotic fluid injected in skin edges

INTERVENTIONS:
Biological: autologous amniotic fluid — 10 cc of amniotic fluid aspirated after opening uterine incision in cesarean section, then Injected in edges of skin before closure
  Arms: cases
Other: No amniotic fluid injected in skin edges — conventional closure of skin
  Arms: control

SUMMARY:
The goal of this randomized controlled trial is to investigate the effect of injection of autologous amniotic fluid in the healing of the scar of cesarean section among high-risk population. Investigator's aim is to know : quality of wound healing, rate of infection and time needed for complete healing. Participants will be divided into two groups. All participants will undergo cesarean section. We will inject autologous amniotic fluid in the edges of the wound during skin closure in half of the participants. Wound healing will be assessed at 1st, 2nd and 6th week postoperatively.

DETAILED DESCRIPTION:
After surgery, participants will be observed along 6 weeks (at 1, 2 and 6 weeks intervals) and scars will be assessed regarding color, thickness, pliability and presence of exudate.

ELIGIBILITY:
Inclusion Criteria:

* Age > 30 years old.
* Anemic patients
* Maternal chronic disease e.g., Diabetes and Hypertension
* BMI of > 25 Kg/m2.
* Underwent previous CS.

Exclusion Criteria:

* Rupture of membrane.
* No previous section.
* Anhydraminos.
* Congenital malformation of the fetus.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Quality of wound healing | 1,2,6 weeks postoperative
  Scars will be assessed objectively regarding Color, Thickness, Pliability, Exudate in participants and controls

CONTACTS AND LOCATIONS:
Locations (1):
- kasr Al Aini, Faculty of Medicine, Cairo University, Cairo, Old Cairo, Egypt